### STUDY PROTOCOL

### **Protocol Number**

IC-201

FDA IND Number: 127083

## **Protocol Title**

Pilot Study Evaluating the Efficacy of Certolizumab Pegol for Interstitial Cystitis

### **Date**

November 5, 2015

### **Principal Investigator**

Philip C. Bosch, MD, Urologist Email: <a href="mailto:pboschmd@gmail.com">pboschmd@gmail.com</a>

pbosch@ucsd.edu

Cell phone: (760) 518-2421

### Official Name

IC Study, LLC 651 E. Pennsylvania Ave. Ste. 201 Escondido, CA 92025 (760) 743-0532

Email: icbpsstudy@gmail.com

Web site: <a href="ICStudy.net">ICStudy.net</a>

### **Recruitment and Study Sites**

Philip C. Bosch, MD 651 E. Pennsylvania Ave. Ste. 201 Escondido, CA 92025 (760) 743-3135

Department of Urology University of California, San Diego Medical Center 200 West Arbor Drive San Diego, CA USA 92103

### **Laboratory**

Quest Diagnostics 8410 Fallbrook Ave. West Hills, CA 91304 800 287-4309

# **Institutional Review Board**

Aspire IRB

Protocol: IC-201 Approval: 7/24/2015 11491 Woodside Ave. Santee, CA 92071 619 469-0108

### Purpose and Study Background

Interstitial cystitis/ bladder pain syndrome (IC/BPS) is a chronic, debilitating bladder disease characterized by suprapubic pressure or pain accompanied by urinary frequency and urgency, in the absence of an identifiable cause. Population based studies have demonstrated a prevalence rate of 3 to 12 percent among women and 2 to 4 percent for men. The symptoms of IC/BPS result in a poor quality of life with sleep dysfunction, sexual dysfunction, depression, anxiety, and stress.

The pathogenesis of IC/BPS is undefined. Treatments of IC/BPS have been empirical and inadequate. Narcotics are the most commonly prescribed medication. The direct cost of medical care for IC/BPS patients is > \$11,000 per year. There are also the indirect costs to society including work absenteeism and decreased productivity. Investigation of novel therapies is needed.

IC/BPS has been postulated to be one of the autoimmune diseases. Like autoimmune diseases, IC/BPS affects more women than men. Infection and stress worsen both conditions. Pregnancy improves symptoms for both IC/BPS and autoimmune diseases. There is a clinical concordance of IC/BPS with other established autoimmune diseases. IC/BPS as an autoimmune disease is not a new theory. In 1938 Fister recognized the clinical and histopathologic similarities between IC/BPS and lupus erythematosus. In the 1980 review article, Oravisto viewed IC/BPS as an autoimmune disease due to the very chronic course of the disease, the absence of infection, the pathological findings, the common occurrence of antinuclear antibodies, and the response to certain modalities of treatment. In Immunosuppressive drugs including methotrexate, prednisone, and cyclosporine A, routinely used to treat autoimmune diseases, have shown efficacy in selected IC/BPS patients. There are more than 80 different documented autoimmune diseases affecting every organ and tissue in the body. IC/BPS may be the autoimmune disease of the bladder.

Selective release of tumor necrosis factor-alpha (TNF $\alpha$ ) by mast cells (MC) plays a central role in the pathogenesis and pathophysiology of IC/BPS. Bladder biopsies of patients with IC demonstrate increase numbers of MC. A selective release or degranulation of vasoactive and proinflammatory mediators by MC, a process called "activation", may explain IC/BPS pathogenesis. MC activation elicits an inflammatory response in urothelial cell IC/BPS models with secreted product TNF $\alpha$  playing a central role. Inflammation in experimental IC/BPS was mediated by TNF $\alpha$ . Drugs that inhibited TNF $\alpha$  decreased this experimental IC/BPS bladder inflammation. Interruption of mast cell activation, with a decrease expression of TNF $\alpha$ , inhibited bladder inflammation in an autoimmune cystitis model.

Elevated levels of TNFα in urine, serum, and tissue were found in patients with IC/BPS. TNFα, a proinflammatory cytokine released by immune cells, is central to the acute and chronic inflammation in autoimmune diseases.  $^{32,33}$  Patients with clinically diagnosed IC/BPS, but no glomerulations observed with cystoscopy under anesthesia after hydrodistention, had elevated levels of TNFα in urine or bladder wash fluid.  $^{34}$  However, patients with clinically diagnosed IC/BPS, but did have glomerulations observed with cystoscopy under anesthesia after hydrodistention, did not have elevated levels of TNFα in urine or bladder wash fluid compared to controls. Interestingly, cystoscopic findings were not felt to identify distinct subgroups of patients with IC/BPS symptoms. TNFα was upregulated in urine of patients with overactive bladder a syndrome that has been considered a milder form of IC/BPS. Serum levels of TNFα were significantly higher in patients with IC/BPS. Tissue levels of TNFα were significantly elevated in women with vulvar vestibulitis. Vulvar vestibulitis, also known as vulvodynia is part of the symptom complex in women with IC/BPS. TNFα is highly expressed in bladder urothelium tissue of patients with ulcerative IC/BPS and was suggested to be the causative etiology of IC/BPS.

I recently completed a study (ClinicalTrials.gov Identifier NCT01295814) "A Randomized, Double-Blind, Placebo Controlled Trial of Adalimumab in the Treatment of Interstitial Cystitis/Bladder Pain Syndrome". Adalimumab is one of several biological agents that are known as TNFα antagonists or TNFα blocking agents. Adalimumab is a recombinant, fully human, monoclonal antibody that neutralizes human TNFα. In this study adalimumab treatment demonstrated a statistically significant improvement in outcome measures compared to baseline in patients with moderate to severe IC/BPS. However, adalimumab failed to demonstrate positive proof of concept compared to placebo due to a significant placebo effect. This confounding result was evaluated and analyzed in my paper "Examination of the Significant Placebo Effect in the Treatment of Interstitial Cystitis/ Bladder Pain Syndrome". The

conclusions of this paper were that this greater "placebo effect" represented the benefits of advice, support, education, and behavior modification programs. The recommendation was that physicians should review standard advice with all IC/BPS patients before starting medical therapy or clinical trials. Future studies should include a washout period after subjects receive standard IC/BPS advice. Only those patients who do not improve with standard IC advice and therapy would be participants in clinical trials.

Current understanding of the TNF $\alpha$  blocking agents recognizes differences in each of their mechanism of action and clinical experience. Adalimumab may not theoretically be the best TNF $\alpha$  blocking agent for the treatment of IC/BPS. Adalimumab mediates complement-dependent cytotoxicity and antibody-dependent cell-mediated cytotoxicity. Adalimumab increases the proportion of cells undergoing apoptosis and the level of granulocyte degranulation. <sup>44</sup> This may not be therapeutically beneficial as IC/BPS histologically demonstrates a pancystitis with mast cell infiltration. <sup>45</sup> A total degranulation of these inflammatory cells with the release of histamine, cytokines, and proteolytic enzymes, typical of an anaphylactic reaction, may exacerbate bladder inflammation.

Certolizumab pegol (Cimzia) has some advantages over other TNF $\alpha$  blocking agents for the treatment of IC/BPS including better distribution in inflamed tissue<sup>46</sup>, development of low levels of neutralizing autoantibodies<sup>47</sup>, greater affinity to TNF $\alpha$ <sup>48</sup>, and efficacy when used in monotherapy<sup>49</sup>. Patients with rheumatoid arthritis treated with certolizumab pegol demonstrated a rapid clinical response, often within 2 weeks. Certolizumab pegol inhibits cytokine production.<sup>44</sup> Certolizumab pegol has a unique mechanism of action that should be beneficial in the treatment of IC/BPS in that it has no complement-dependant cytotoxicity and antibody-dependant cell-mediated cytotoxicity.<sup>44,50</sup> IC/BPS histologically demonstrates a pancystitis with mast cell infiltration.<sup>45</sup> The polyethylene glycol moiety of certolizumab pegol inhibits mast cell degranulation.<sup>51</sup> TNF $\alpha$  blocking agents that do not cause cytolysis and prevents degranulation of these inflammatory cells should be therapeutically beneficial in the treatment of IC/BPS.

Most trials in IC/BPS use a patient-reported global response assessment (GRA) such as "Compared to when you began this trial, how would you rate your IC symptoms now?" as the primary endpoint. The O'Leary-Sant Interstitial Cystitis Symptom Index and Problem Index (OSPI) questionnaire evaluates overall symptoms in IC/BPS patients. The OSPI results confirm the clinical diagnosis of IC/BPS and establish the severity of the participants IC/BPS baseline symptoms. The Interstitial Cystitis Symptom Index (ICSI) is one of the two O'Leary-Sant Interstitial Cystitis Symptom and Problem Indexes. ICSI has been validated as a reliable

and responsive measure of changes in IC/BPS symptoms.<sup>53,55</sup> ICSI is recommended as an endpoint in IC clinical trials.

Research has searched unsuccessfully for an inflammatory urine biomarker for the diagnosis of IC/BPS. However, Felson<sup>34</sup> demonstrated elevated urine TNF $\alpha$  levels measured by ELISA in patients with IC/BPS compared to controls. It would be interesting to measure urine TNF $\alpha$  levels with modern techniques in IC/BPS patients and see if those levels go down with certolizumab pegol treatment.

The FDA asked for more outcome measures so ICPI and numeric rating scale for pain and urgency was added. They asked for monitoring of patient with outcome data to week 18. We also agreed to change the potential total number of patients from 44 to 42 as this would maintain the 2:1 study medication ratio.

| <b>Condition</b> | <u>Intervention</u> | <b>Phase</b> |
|---|---|---|
| Cystitis, Interstitial | Biological: Certolizumab pegol (Cimzia) | Phase III |
| Bladder Pain Syndrome | Other: Placebo | |

Study Type: Interventional

Study Design: Randomized, Double-Blind, Placebo Controlled Treatment, Efficacy Study

### **Primary Outcome Measures**

The primary endpoint is improvement in global response assessment (GRA) at week 2

### **Secondary Outcome Measures**

Improvement in GRA at week 4, 10, and 18

Improvement in the Interstitial Cystitis Symptom Index (ICSI) Interstitial Cystitis Problem Index (ICPI) from baseline to week 2, 4, 10, and 18

11-point numeric pain and urgency scale at baseline, week 2, 4, 10, and 18

Midstream first void urine specimen level of TNF $\alpha$  normalized to urinary creatinine, at week 2,

4, 10, and 18 compared to baseline levels

Adverse events from time of Screening through the last clinic and phone call visit

# **Estimated enrollment** 42 patients

After subjective evaluation of efficacy and safety in the initial 30 patients, the total study sample size will be 42 study patients.

Previous IC/BPS studies demonstrated an approximate 20% placebo response rate. Monotherapy response rate of certolizumab pegol in rheumatoid arthritis was 45%. To achieve an 80% power using 2:1 randomization and a 2-sided p = .05 a minimum of 39 subjects was required. The sample size was increased by 3 subjects to account for potential participant withdrawals.

| <u>Arms</u> | Assigned Intervention |
|---|---|
| Group 1:<br>Experimental | Biological: Certolizumab pegol (Cimzia) 400 mg pre-filled syringe loading dose given subcutaneously at week 0, 2, and 4 followed by a maintenance dose at week 8 |
| Group 2: Placebo<br>Comparator | Placebo: given subcutaneously at week 0, 2, 4, and week 8 |

# **Eligibility**

Ages Eligible for Study: 18-65

Genders Eligible for Study: Female

### **Inclusion Criteria**:

- 1. A diagnosis of IC/BPS defined based on AUA guidelines as the following: an unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms of more than 6 months duration, in the absence of infection or identifiable causes, documented history or patient reported.
- 2. Only those patients with moderate to severe IC/BPS will be included in the study.
- 3. Able to provide informed consent to participate in the study and comply with study requirements
- 4. Able to provide written authorization for use and release of health and research study information
- 5. Written documentation of being provided California's Experimental Subject's Bill of Rights
- 6. Females ≥18 and ≤ 65 years of age previously diagnosed with interstitial cystitis/ bladder pain syndrome (IC/BPS) for a duration of greater than 6 months
- 7. Female patients of child-bearing potential must have a negative serum pregnancy test at Screening and use birth control while in the study.
- 8. O'Leary-Sant Interstitial Cystitis Symptom and Problem Indexes (OSPI) score ≥ 18
- 9. No history of any cancer.
- 10. No bacterial cystitis in previous 1 month
- 11. No active herpes in previous 3 months
- 12. Never treated with cyclophosphamide
- 13. No neurogenic bladder dysfunction (due to a spinal cord injury, stroke, Parkinson's disease, multiple sclerosis, spina bifida or diabetic cystopathy)
- 14. Absence of bladder, ureteral or urethral calculi for previous 3 months

#### **Exclusion criteria:**

- 1. Symptoms are relieved at one month reevaluation visit after receiving IC/BPS behavior modification advice at screening visit.
- 2. Symptoms are relieved by antimicrobials, antibiotics, or other medications for IC/BPS
- 3. Pregnant women, lactating mothers, nursing mothers, women suspected of being pregnant and woman who plan to be pregnant during the course of the clinical trial
- 4. Males
- 5. Patients with inadequate renal, hepatic, or cardiac function
- 6. Patients with history of gross hematuria within 2 years.
- 7. Patients with the following medical history: Lower urinary tract anatomical anomaly, pelvic radiotherapy, or active genital herpes
- 8. Patients with a history of tuberculosis (TB), recent exposure to TB, or recent travel to TB endemic regions. Patients should have a recent negative PPD (or negative CXR) prior to receiving treatment.
- 9. Patients who have undergone cystoscopy under anesthesia with bladder biopsy, hydrodistension, or fulguration of Hunner's ulcer within 3 months
- 10. Patients taking the following treatments for interstitial cystitis at Screening: Intravesical BCG, corticosteroid therapy, cyclosporine, or TNF-alpha inhibitors.
- 11. Patients with a history of receiving live vaccine including Flumist® influenza vaccine in the past 3 months.
- 12. Patients with a history of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG-fusion protein.

- 13. Patients with a history of alcohol, analgesic or drug abuse within 2 years of Screening.
- 14. Patients with a history of any cancer.
- 15. Patients with a history of active Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus (HIV) infection, or who are known carriers (Hepatitis B).
- 16. Patients with a history of invasive fungal infections, recent travel to regions endemic for the following invasive fungal infections: San Joaquin Fever, aspergillosis, histoplasmosis, candidiasis, coccidiodomycosis, blastomycosis, and pneumocystosis.
- 17. Patients with a history of diabetes mellitus.
- 18. Patients with a history of a neurologic disease included but not limited to central demyelinating diseases, including multiple sclerosis; and a history of peripheral demyelinating disease, including Guillain-Barre syndrome.
- 19. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.

### **Study Design**

Patients enter a one month Screening period to assess inclusion/exclusion criteria, sign informed consent, and determine study eligibility. At the initial screening visit, patients will be instructed in behavior modification techniques to improve IC/BPS symptoms. <sup>43</sup> Patients are reassessed at least one month later for inclusion/exclusion criteria and determine study eligibility. Patients who do not improve with standard IC/BPS advice and pass clinical and laboratory screening can be participants in the study. Baseline evaluation of the included patients will be done with the O'Leary-Sant Interstitial Cystitis Symptom Index and Problem Index (OSPI). At the baseline visit (week 0), all eligible IC/BPS patients will be randomized in a blinded fashion to receive in a 2:1 ratio either SQ certolizumab pegol 400mg or SQ placebo at weeks 0, 2, 4 followed by a maintenance dose at 8 weeks. The length of the study will be 18 weeks. The effectiveness of certolizumab pegol will be assessed at week 2, 4, 10, and 18 using GRA, ICSI, ICPI, and the numeric pain and urgency scale. After subjective evaluation of efficacy and safety in the initial 30 patients, the total study sample size will be 42 study patients.

A midstream urine will be collected at baseline and weeks 2, 4, 10, and 18 from all participants. Quest Diagnostics Nichols Institute, San Juan Capistrano, CA or similar lab will perform an ELISA TNFα and creatinine levels on these samples.

Pilot Study Evaluating the Efficacy of CZP for Interstitial Cystitis Study Flow Chart



# **Trial Schedule**

| | Screen | >One Month<br>Reevaluation | Baseline | Visit<br>1 | Visits 2, 3 | Visit 4 | Phone<br>Follow-<br>up <sup>6</sup> | Phone<br>Follow-<br>up <sup>6</sup> |
|---|---|---|---|---|---|---|---|---|
| Study Day | -37 | -7 | 0 | 14 | 28,56 | 70 | 98 | 126 |
| Study Week | -5 | -1 | 0 | 2 | 4,8 | 10 | 14 | 18 |
| Study | | | | | | | | |
| procedures: | | | | | | | | |
| Obtain Informed<br>Consent | X | | | | | | | |
| Medical History | X | | | | | | | |
| Medication<br>Review | X | X | X | X | X | X | | |
| Vitals <sup>1</sup> | X | X | X | X | X | X | | |
| Physical Exam | X | | | | | | | |
| OSPI <sup>2</sup> | X | X | | | | | | |
| anti-HCV, HBsAG | | X | | | | | | |
| PPD | | X | | | | | | X |
| CBC | | | | | | X | | X |
| Urinalysis | X | X | X | X | X | X | | |
| Urine Culture | | X | X | X | X | X | | |
| Urine Pregnancy<br>Test | | X | | | | | | |
| Eligibility<br>Assessment | X | X | | | | | | |
| Dispense Study<br>Drug | | | X | X | X | | | |
| Injection Site<br>Evaluation <sup>3</sup> | | | X | X | X | | | |
| Adverse Events | | | X | X | X | X | X | X |
| GRA <sup>4</sup> | | | | X | X | X | | X |
| ICSI, ICPI <sup>5</sup> | | | | X | X | X | | X |
| Numeric scale of pain and urgency | X | X | X | X | X | X | | X |

- 1. Height, weight, blood pressure, pulse, temperature
- 2. O'Leary-Sant Interstitial Cystitis Symptom Index and Problem Index
- 3. Monitor subjects for systemic and local hypersensitivity reactions for one hour after injection

- 4. Global response assessment
- 5. Interstitial Cystitis Symptom Index, Interstitial Cystitis Problem Index
- 6. In-office visit if determined to be clinically necessary

### **Statistical Analysis**

All statistical summaries and 2-sample t-tests were performed using the Data Desk® version 6.3. Comparison of these changes between treatment groups are also shown as 95% confidence intervals (CI). The chi-square test or Fisher's exact test was applied to analyze baseline demographics, improvement with GRA treatment responders, and the proportion of patients with a reduction from baseline of 30% or greater in their pain intensity score between treatment groups.

### **Safety Evaluation**

Patients will be assessed at office visits and by continuous availability by phone for adverse events. Adverse effects may include rhinitis, headache, rash, pruritus, injection site reaction, infections, tuberculosis, cancer, and demyelinating diseases.

#### **Stopping Criteria for Adverse Events**

#### **Serious infections:**

These include TB and infections caused by viruses, fungi, or bacteria. Symptoms related to TB include cough, low-grade fever, weight loss, or loss of body fat and muscle.

### Allergic reactions:

Signs of a serious allergic reaction include skin rash, a swollen face, or trouble breathing.

### **Nervous system problems:**

Signs and symptoms include numbness or tingling, problems with your vision, weakness in your arms or legs, and dizziness.

# **Blood problems**:

Symptoms include a fever that does not go away, bruising or bleeding very easily, or looking very pale.

# New heart failure or worsening of heart failure you already have:

Symptoms include shortness of breath or swelling of your ankles or feet, or sudden weight gain.

# Immune reactions including a lupus-like syndrome:

Symptoms include chest discomfort or pain that does not go away, shortness of breath, joint pain, or rash on your cheeks or arms that gets worse in the sun.

### References

- 1. Simon LJ, Landis JR, Erickson DR et al: The Interstitial Cystitis Data Base Study: concepts and preliminary baseline descriptive statistics. Urology 1997; **49(Suppl 5A):** 64.
- 2. van de Merwe JP, Nordling J, Bouchelouche K et al: Diagnostic criteria, classification, and nomenclature for painful bladder syndrome/interstitial cystitis: an ESSIC proposal. Eur Urol 2008; **53:** 60.
- 3. Hanno P, Lin A, Nordling J et al: Bladder pain syndrome committee of the international consultation on incontinence. Neurourol Urodyn 2010; **29:** 191.
- 4. Clemens JQ, Meenan RT, Rosetti M et al: Prevalence of interstitial cystitis symptoms in a managed care population. J Urol 2005; **174:** 576.
- 5. Rosenberg MT and Hazzard M: Prevalence of interstitial cystitis symptoms in women: a population based study in the primary care office. J Urol 2005; **174:** 2231.
- 6. Berry SH, Eliott MN, Suttorp M et al: Prevalence of symptoms of bladder pain syndrome/interstitial cystitis among adult females in the United States. J Urol 2011; **186:** 540.
- 7. Michael YL, Kawachi I, Stampfer MJ et al: Quality of life among women with interstitial cystitis. J Urol 2000; **164:** 423.
- 8. Rothrock NE, Lutgendorf SK, Hoffman A et al: Depressive symptoms and quality of life in patients with interstitial cystitis. J Urol 2002; **167:** 1763.
- 9. Nickel JC, Tripp DA, Pontari M et al: Psychosocial phenotyping in women with interstitial cystitis/painful bladder syndrome: a case control study. J Urol 2010; **183:** 167.
- 10. Propert KJ, Schaeffer AJ, Brensinger CM et al: A prospective study of interstitial cystitis: results of longitudinal followup of the interstitial cystitis data base cohort. The Interstitial Cystitis Data Base Study Group. J Urol 2000; **163:** 1434.
- 11. Phatak S, and Foster HE: The management of interstitial cystitis: an update. Nat Clin Pract 2006; **3(1):** 45.
- 12. Dimitrakov J, Kroenke K, Steers WD et al: Pharmacologic management of painful bladder syndrome/interstitial cystitis A systematic review. Arch Intern Med 2007; **167(18):** 1922.
- 13. Anger JT, Zabihi N, Clemens JQ et al: Treatment choices, duration, and cost in patients with interstitial cystitis and painful bladder syndrome. Int Urogynecol J 2011; **22:** 395.
- 14. Robinson R: The economic burden of interstitial cystitis and painful bladder syndrome. J Urol 2011; **185(4S):** e129.
- 15. Alagiri M, Chottiner S, Ratner V et al: Interstitial cystitis: unexplained associations with other chronic disease and pain syndromes. Urology 1997; **49(5A):** 52.

- 16. Fister GM: Similarity of interstitial cystitis to lupus erythematosus. J Urol 1938; 40: 37.
- 17. Oravisto KJ: Interstitial cystitis as an autoimmune disease. A review. Eur Urol 1980; **6:** 10.
- 18. Moran PA, Dwyer PL, Carey MP et al: Oral methotrexate in the management of refractory interstitial cystitis. Aust N Z Obstet Gynaecol 1999; **39:** 468.
- 19. Soucy F and Gregoire M: Efficacy of prednisone for severe refractory ulcerative interstitial cystitis. J Urol 2005; **173:** 841.
- 20. Forrest JB, Payne CK, Erickson DR: Cyclosporine A for refractory interstitial cystitis/bladder pain syndrome: Experience at 3 tertiary centers. J Urol 2012; **188:** 1186.
- 21. Larsen S, Thompson SA, Hald T et al: Mast cells in interstitial cystitis. Brit J Urol 1982; **54:** 283.
- 22. Feltis JT, Perez-Marrero R, and Emerson LE: Increased mast cells of the bladder in suspected cases of interstitial cystitis: a possible disease marker. J Urol 1987; **138:** 42.
- 23. Theoharides TC, Sant GR, el-Mansoury M et al: Activation of bladder mast cells in interstitial cystitis: a light and electron microscopic study. J Urol 1995; **153:** 629.
- 24. Letourneau R, Pang X, Sant GR et al: Intragranular activation of bladder mast cells and their association with nerve processes in interstitial cystitis. Br J Urol 1996; 77: 41.
- 25. Theoharides TC, Kempuraj D, and Sant GR: Mast cell involvement in interstitial cystitis: a review of human and experimental evidence. Urology 2001; **57** (**suppl 6A**): 47.
- 26. Batler RA, Sengupta S, Forrestal SG et al: Mast cell activation triggers a urothelial inflammatory response mediated by tumor necrosis factor-α. J Urol 2002; **168:** 819.
- 27. Chen MC, Blunt LW, Pins MR et al: Tumor necrosis factor promotes differential trafficking of bladder mast cells in neurogenic cystitis. J Urol 2006; **175:** 754.
- 28. Gonzales RR, Fong T, Belmar N et al: Modulating bladder neuro-inflammation: RDP58, a novel anti-inflammatory peptide, decreases inflammation and nerve growth factor production in experimental cystitis. J Urol 2005; **173:** 630.
- 29. Boucher W, Kempuraj D, Cao J et al: Intravesical suplatast tosilate (IPD-1151T) inhibits experimental bladder inflammation. J Urol 2007; **177:** 1186.
- 30. Boucher W, Stern JM, Kotsinyan V et al: Intravesical nanocrystalline silver decreases experimental bladder inflammation. J Urol 2008; **179:** 1598.
- 31. Liu WJ and Luo Y: Interruption of mast cell function effectively inhibits bladder inflammation in an autoimmune cystitis model. J Urol 2008; **179** (suppl 4): 62.
- 32. Feldmann M: Development of anti-TNF therapy for rheumatoid arthritis. Nat Rev Immunol 2002; **2:** 364.

- 33. Tracey D, Klareskog L, Sasso EH et al: Tumor necrosis factor antagonist mechanisms of action: a comprehensive review. Pharmacol Ther 2008; **117:** 244.
- 34. Felsen D, Frye S, Trimble LA et al: Inflammatory mediator profile in urine and bladder wash fluid of patients with interstitial cystitis. J Urol 1994; **152:** 355.
- 35. Erickson DR, Tomaszewski JE, Kunselman AR et al: Do the National Institute of Diabetes and Digestive and Kidney Diseases cystoscopic criteria associate with other clinical and objective features of interstitial cystitis. J Urol 2005; **173:** 93.
- 36. Ghoniem G, Faruqui N, Elmissiry M et al: Differential profile analysis of urinary cytokines in patients with overactive bladder. Int Urogynecol J 2011; **22:** 953.
- 37. MacDiarmid SA and Sand PK: Diagnosis of interstitial cystitis/painful bladder syndrome in patients with overactive bladder symptoms. Rev Urol 2007; **9(1):** 9.
- 38. Jiang YH, Peng CH, Liu HT et al: Increased pro-inflammatory cytokines, C-reactive protein and nerve growth factor expressions in serum of patients with interstitial cystitis/bladder pain syndrome. PLoS ONE 2013: **8(10):** e76779.
- 39. Foster DC and Hasday JD: Elevated tissue levels of interleukin-1β and tumor necrosis factor- α in vulvar vestibulitis. Obstet Gynecol 1997; **89(2):** 291.
- 40. Gardella B, Porru D, Nappi RE et al: Interstitial cystitis is associated with vulvodynia and sexual dysfunction- a case-control study. J Sex Med 2011; **8(6):** 1726.
- 41. Ogawa T, Homma T, Igawa Y et al: CXCR3 binding chemokine and TNFSF14 over expression in bladder urothelium of patients with ulcerative interstitial cystitis. J Urol 2010; **183**: 1206.
- 42. Bosch PC: A randomized, double-blind, placebo controlled trial of adalimumab in the treatment of interstitial cystitis/bladder pain syndrome. J Urol 2014; **191:** 77.
- 43. Bosch PC: Examination of the significant placebo effect in the treatment of interstitial cystitis/ bladder pain syndrome. Urology 2014; **84:** 321.
- 44. Nesbitt A, Fossati G, Bergin M et al: Mechanism of action of certolizumab pegol (CDP870): in vitro comparison with other anti-tumor necrosis factor α agents. Inflamm Bowel Dis 2007; 13
  (II): 1323.
- 45. Larsen S, Thompson SA, Hald T et al: Mast cells in interstitial cystitis. Brit J Urol 1982; **54:** 283.
- 46. Marenzana M, Eddleston A, Vulger A et al: Differential distribution of a pegylated Fab' into inflamed versus normal tissue compared with an IGG in arthritis and colitis models (abstract). Ann Rheum Dis 2010; **69(suppl 2):** A61.
- 47. Schreiber S, Khaliq-Kareemi M, Lawrence IC et al: Maintenance therapy with certolizumab pegol for Crohn's Disease. NEJM 2007; **357:** 239.

- 48. Nesbitt AM and Henry AJ: High affinity and potency of the pegylated Fab fragment CDP870. Am J Gastroenterol 2004; **99**; S253.
- 49. Fleischmann R, Vencovsky J, and van Vollenhoven RF: Efficacy and safety of certolizumab pegol monotherapy every 4 weeks in patients with rheumatoid arthritis failing previous disease-modifying antirheumatic therapy: the FAST4WARD study. Ann Rheum Dis 2009; **68(6):** 805.
- 50. Bourne T, Fossati G, and Nesbitt A: A pegylated Fab' fragment against tumor necrosis factor for the treatment of Crohn's Disease: exploring a new mechanism of action. BioDrugs 2008; **22:** 331.
- 51. Lamour S, Bracher M, and Nesbitt A: The PEG component of certolizumab pegol inhibits degranulation by stimulated mast cells (abstract). Arthritis Rheum 2009; **60(suppl 10):** 44.
- 52. Sant GR, Propert KJ, Hanno PM et al: A pilot clinical trial of oral pentosan polysulfate and oral hydroxyzine in patients with interstitial cystitis. J Urol 2003; **170**: 810.
- 53. Propert KJ, Mayer RD, Wang Y et al: Responsiveness of symptom scales for interstitial cystitis. Urology 2006; **67:** 55.
- 54. O'Leary MP, Sant GR, Fowler FJ et al: The interstitial cystitis symptom index and problem index. Urology 1997; **49** (suppl 5A): 58.
- 55. Lubeck DP, Whitmore K, Sant GR et al: Psychometric validation of the O'Leary-Sant interstitial cystitis symptom index in a clinical trial of pentosan polysulfate sodium. Urology 2001; **57(Suppl 6A):** 62.
- 56. Hwang P, Auclair B, Beechinor D, Diment M, Einarson TR. Efficacy of pentosan polysulfate in the treatment of interstitial cystitis: a meta-analysis. Urology 1997;50:39.